CLINICAL TRIAL: NCT05662995
Title: Point-of-care Ultrasound Abnormalities in Early Onset Preeclampsia - Prevalence and Association Between Pulmonary Interstitial Syndrome and Cardiac Dysfunction, Brain Natriuretic Peptide, and Serum Albumin
Brief Title: Point-of-care Ultrasound Abnormalities in Early Onset Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Dyer, Professor Robert Dyer, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: POCUS in early preeclampsia
Record Dates: First submitted 2022-11-22; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Preeclampsia; Pulmonary Edema; Cardiac Function
MeSH Terms: conditions — Pre-Eclampsia; Pulmonary Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung- and cardiac ultrasound, as well as optic nerve sheath diameter. (Experimental): An ultrasound examination (approximately 25-30 minutes in duration) will be performed at the time of venous blood sampling on admission. The examination will consist of an assessment of systolic and diastolic function, lung ultrasound, and measurement of the optic nerve sheath diameter
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound will be performed with the patient in supine position (with or without left uterine displacement, depending on clinical circumstances). A phased-array transducer will be used for lung ultrasound and will be used for the assessment of B-lines, which arise from the pleural line and extend to the bottom of the screen and move with the sliding lung

SUMMARY:
The study is planned to describe the prevalence and severity of cardiac, lung and optic-nerve sheath diameter (ONSD) ultrasound abnormalities in women with early onset preeclampsia with severe features. These findings will be compared with point-of-care ultrasound (POCUS) abnormalities demonstrated in our recent study on late onset preeclampsia. The primary aim of the current study will be to examine the association between pulmonary interstitial edema (PIS), as identified by lung ultrasound, and cardiac dysfunction on echocardiography, and brain natriuretic peptide (BNP), in early onset preeclampsia, after comprehensive echocardiographic assessment. The secondary aims are to assess ONSD, and to explore the association between PIS or ONSD and serum albumin. A further secondary aim will be to explore the association between POCUS abnormalities and cardiotocography abnormalities and early delivery.

DETAILED DESCRIPTION:
Preeclampsia (PE) remains a leading cause of maternal morbidity and mortality, in both high-, low and-middle-income countries. It is a complex, multisystem disease which, in its severe form, affects the cardiovascular, renal, hepatic, neurological and haematological systems. The University of Cape Town-associated medical institutions alone were responsible for the treatment of approximately 800 women in 2019, who were classified as having PE with severe features. Recent studies have demonstrated novel markers of severity of PE, including point-of-care ultrasound (POCUS), acid-base changes secondary to low serum albumin, and brain natriuretic peptide (BNP). A study conducted at Mowbray Maternity Hospital in Cape Town, South Africa, showed that approximately 59% of women had an abnormality shown by POCUS; 24% had elevated lung water (pulmonary interstitial syndrome [PIS]). These findings could serve as non-invasive markers of disease severity, and thus may be used to predict maternal and fetal outcome in preeclamptic women. POCUS is playing an increasing role in perioperative diagnosis, and newer, less expensive devices are continuously being developed. These will in all likelihood play an important role in South Africa in the near future. In a recent trial performed at the University of Cape Town, a comprehensive acid-base analysis in women with PE with severe features demonstrated significant abnormalities in independent acid-base determinants. In addition, strong indications were found that changes in acid-base status following a decrease in serum albumin are more pronounced in early onset PE, and may be associated with urgent delivery. In other clinical arenas in critically ill patients, low serum albumin is associated with increased lung water, increased intracranial pressure, and outcome. The study team hypothesised that similar associations might be found in women with late onset preeclampsia with severe features. Using POCUS, it was found that there was no association between serum albumin level and PIS or optic nerve sheath diameter (ONSD). PIS was however associated with cardiac dysfunction, as was BNP. This study is planned to describe the prevalence of pulmonary (PIS), cardiac and optic nerve sheath abnormalities found on ultrasound in women diagnosed with early onset PE with severe features. In a recent study on POCUS findings in late onset preeclampsia, the absence of PIS may exclude raised LVEDP. As a consequence, the primary aim of the current study is to examine the association between PIS, as identified by lung ultrasound and cardiac dysfunction on echocardiography, and BNP, in early onset PE. For this purpose, a comprehensive echocardiographic assessment will be performed. The secondary aims are to explore the association between PIS or ONSD and serum albumin. These findings will be compared with POCUS abnormalities demonstrated in our recent study on late onset PE. In addition, the association will be explored between POCUS abnormalities and CTG abnormalities and early delivery. Using a prospective observational cohort design, patients diagnosed with early onset PE with severe features will be enrolled. If agreeable to participate in the study, a venous blood sample will be taken for the measurement of serum BNP and serum albumin level, followed by a 25-30 minute non-invasive lung, cardiac and optic nerve ultrasound examination. The risks posed to the patients involved in this study are minimal. Discomfort may be experienced due to the sampling of blood, however these will be performed as part of the routine blood sampling in patients with PE. All ultrasound interventions are non-invasive. Patients not included in the study will not be disadvantaged in any way, as no treatment interventions are being proposed. All study participants will be clinically managed by the attending obstetrics team and collaborative involvement with the team will ensure current management standards at the Maternity Centre at Groote Schuur Hospital in Cape Town are maintained. Thus, the 25-30 minute ultrasound examination will not interfere with or compromise standard healthcare to recruited study participants. This observational study carries minimal risk and has the potential to fill a major knowledge gap in the role of ultrasound in the anaesthesia care of preeclamptic patients. This should be of significant future benefit in the South African context, where PE is a leading cause of maternal mortality and pulmonary oedema is a main contributor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed and admitted with early onset preeclampsia with severe features

Exclusion Criteria:

1. Body mass index (BMI) > 50 kg/m2
2. Clinical evidence of pulmonary oedema
3. The presence of a non-reassuring fetal heart trace
4. Active labour
5. Chronic pulmonary disease, or acute asthma
6. Collagen disorders
7. Chronic renal or hepatic disease
8. Urinary tract infection
9. Chorioamnionitis
10. Intrauterine fetal death
11. Patients unable to provide informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women.
Enrollment: 60 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The association between pulmonary interstitial syndrome and cardiac dysfunction on echocardiography | 35-40 minutes
  More than 3 B-lines in 2 lung windows bilaterally defines the presence of pulmonary interstitial syndrome.
  Cardiac dysfunction on echocardiography is defined as raised left ventricular end-diastolic pressure as demonstrated on echocardiography.

SECONDARY OUTCOMES:
The association between pulmonary interstitial syndrome or optic nerve sheath diameter, and serum albumin | 35-40 minutes.
  Please see description for outcome 1 for pulmonary interstitial syndrome. Abnormal optic nerve sheath diameter is defined as greater than 5.8 mm. Brain natriuretic peptide and serum albumin are continuous variables.
The prevalence and severity of cardiac, lung and optic nerve sheath diameter abnormalities in women with early onset PE | 35-40 minutes
  Please see definitions as described under Outcome 1 and Outcome 2.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dyer, MBChB, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months following publication.
Access Criteria: Any researchers, and clinicians or healthcare workers continuing care of the participants after the study, as well as the participants themselves.